CLINICAL TRIAL: NCT06094140
Title: NEO-adjuvant Chemo-Immunotherapy in Pancreatic Cancer
Acronym: NEO-IMPACT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: The University of New South Wales (Other); Walter and Eliza Hall Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEO-IMPACT
Record Dates: First submitted 2023-08-07; First posted 2023-10-23 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Resectable; Border-line; Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — durvalumab; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm study, mFOLFIRINOX and durvalumab, neoadjuvant resectable pancreatic cancer. (Experimental): All patients enrolled to this study will receive mFOLFIRINOX, delivered Q2W for 6 cycles and durvalumab delivered Q4W for 3 cycles in the neoadjuvant setting for resectable or borderline resectable pancreatic cancer patients. Patients will then undergo restaging, discussion at MDM and surgical resection where appropriate. Following resection, patients will commence 6 cycles of adjuvant mFOLFIRINOX alone (or gemcitabine-based chemotherapy if deemed by investigator as more appropriate).
  Patients will be followed up on study for 12 months from surgery, or from completion of neoadjuvant
  Interventions: Drug: Durvalumab; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Calcium folinate (leucovorin); Drug: Fluorouracil; Drug: Pegylated G-CSF

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be supplied by AstraZeneca as a 500 mg vial concentrate for solution for infusion. The solution contains 50 mg/mL durvalumab, 26 mM histidine/histidine-hydrochloride, 275 mM trehalose dihydrate, and 0.02% weight/volume (w/v) polysorbate 80; it has a pH of 6.0 and density of 1.054 g/mL. The label-claim volume is 10 mL.
  Durvalumab is a sterile, clear to opalescent, colorless to slightly yellow solution, free from visible particles.
  Investigational product vials are stored at 2°C to 8°C (36°F to 46°F) and must not be frozen. Investigational product must be kept in original packaging until use to prevent prolonged light exposure.
  Other Names: Imfinzi
Drug: Oxaliplatin — 85mg/m2 intravenously on day 1
  Other Names: Eloxatin
Drug: Irinotecan — 150mg/m2 intravenously on day 1
  Other Names: Camptosar; Campto
Drug: Calcium folinate (leucovorin) — 50mg as an intravenous bolus
  Other Names: Folinic acid
Drug: Fluorouracil — 2400mg/m2 by continuous infusion via pump over 46 hours starting on day 1
  Other Names: Adrucil
Drug: Pegylated G-CSF — 6mg by subcutaneous injection to be given on day 3 of each cycle.
  Other Names: Neulasta

SUMMARY:
To determine the safety and tolerability of adding durvalumab to mFOLFIRINOX prior to surgery in patients with resectable or borderline resectable pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Despite curative surgery, pancreatic cancer patients have five-year survival rates of 20%. Adjuvant chemotherapy has improved survival in resected pancreatic cancer patients but only 10-15% are suitable for surgery and 30% of the resected pancreatic cancer patients miss out on adjuvant chemotherapy due to postoperative complications.

Neoadjuvant chemotherapy has improved the resection rates in the patients with non-metastatic pancreatic cancer. There is a growing interest to combine chemotherapy with checkpoint inhibitors to improve disease control in the early stage of pancreas cancer. The investigators propose a pilot study to evaluate the feasibility and safety of combining modified FOLFIRINOX (mFOLFIRINOX) with durvalumab (MEDI4736) in patients with resectable or borderline resectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18 years and older, with cytologically or histologically proven resectable or borderline resectable pancreatic adenocarcinoma as per Australasian Gastro-Intestinal Trials Group (AGITG) consensus guidelines. Those in whom cytology is suspicious for pancreatic adenocarcinoma but not diagnostic may be allowed on study following discussion with the study chair (or their representative).
2. ECOG 0-1
3. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥1.5 × 109 /L
   * Platelet count ≥100× 109/L
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). [This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.]
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional ULN unless;

     o There has been recent biliary drainage in the past 30 days, in which case it must be ≤5 x ULN
   * Measured creatinine clearance (CL) >50 mL/min or Calculated creatinine CL >50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: Males: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL) Females: Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 / 72 x serum creatinine (mg/dL)
4. Study treatment both planned and able to start within 14 days of registration.
5. Body weight >30 kg.
6. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
7. Must have a life expectancy of at least 12 weeks.
8. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to first study treatment.
9. Signed, written informed consent.

Exclusion Criteria:

1. Locally advanced or metastatic pancreatic adenocarcinoma.
2. Neuroendocrine pancreatic carcinoma.
3. Prior treatment for pancreatic cancer including chemotherapy, checkpoint inhibitor or investigational treatments, the exception of a maximum of 1 cycle of neoadjuvant intent mFOLFIRINOX.
4. Participation in another clinical study with an investigational product during the last 30 days.
5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or enrolment occurs during the follow-up period.
6. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia.
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
   3. Any chronic skin condition that does not require systemic therapy.
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
   5. Patients with coeliac disease controlled by diet alone.
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, active infection requiring systemic therapy within 14 days before the first dose of study drug, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
11. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease.
12. History of leptomeningeal carcinomatosis.
13. History of active primary immunodeficiency.
14. Active infection including:

    1. Positive test for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies)
    2. Active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice)
    3. Active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (HBcAb or anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of HBcAb or anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
15. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
    4. For patients enrolling after receipt of 1 cycle of mFOLFIRINOX, steroids given pre and post chemotherapy as part of routine care.
16. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
17. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab.
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
19. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
20. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients receiving at least 80% of planned neoadjuvant treatment. | At completion of neo-adjuvant treatment (at 3 months post enrollment)
  80% of planned neoadjuvant treatment is defined as at least 5 cycles of mFOLFIRINOX and at least 2 of 3 cycles durvalumab. Dose modified cycles count towards received treatment.
  Justification: As a pilot study, this primary objective addresses feasibility. A phase II study assessing use of neoadjuvant FOLFIRINOX in borderline resectable pancreatic cancer patients has previously demonstrated an 80% rate of receipt of all planned neoadjuvant therapy (Murphy et al 2018).

SECONDARY OUTCOMES:
The proportion of patients missing surgery due to significant treatment related adverse events. | Every 2 weeks during neo-adjuvant treatment, at the completion of treatment (at 3 months post enrolment) and 30 to 42 days after the last dose of immunotherapy.
  Address efficacy and safety of patients missing surgery due to significant treatment related adverse events.
Treatment tolerability (Rates of adverse events as per CTCAE v5.0). | Through study completion, an average of 1 year
  Address efficacy and safety of treatment tolerability
R0 resection rate. | Through study completion, an average of 1 year
  Address efficacy and safety of the R0 resection rate.
Pathological complete response rate. | Through study completion, an average of 1 year
  Address efficacy and safety of the pathological complete response rate.
Objective response rate. | Through study completion, an average of 1 year
  Address efficacy and safety of the objective response rate.

OTHER OUTCOMES:
To monitor the change in microbiome during neoadjuvant therapy. | At baseline, at end of neoadjuvant treatment (within 2 weeks of last dose) and post-operatively (14-42 days post surgery, prior to commencement of adjuvant treatment)
  Exploratory Objective - Collection of stool samples, oral swabs and tumour tissue to analyse microbiome changes during therapy.
Analysis of tumour tissue (baseline and surgical resection) for molecular changes and gene expression profile. | Through study completion, an average of 1 year
  Exploratory Objective - Immunohistochemistry of immune markers and Fluorescent In-situ Hybridisation to detect tissue localisation of the microbes.

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Chantrill, Professor, Study Chair — AGITG
Locations (3):
- Australia (3):
  - GenesisCare North Shore, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Warringal Private Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No